CLINICAL TRIAL: NCT05723900
Title: Comparative Evaluation of Pulp Response to Castor Oil Versus Formocresol as Pulpotomy Medicaments in Primary Teeth :An in Vivo Study
Brief Title: Evaluation of Pulp Response to Castor Oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Shimaa Hadwa, Lecturer in pediatric dentistry department faculty of dentistry tanta university, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #R-PED-10-22-6,
Record Dates: First submitted 2023-01-22; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2022-10

CONDITIONS: Pulp Response to Castor Oil
MeSH Terms: interventions — Castor Oil; formocresol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Castor oil (Experimental): Castor oil applied to one side of the selected primary canine
  Interventions: Drug: Castor oil
- Formocresol (Experimental): Formocresol applied to other side
  Interventions: Drug: Formocresol

INTERVENTIONS:
Drug: Castor oil — Procedure :pulpotomy procedure and histological evaluation. A sample of sixty two primary teeth from thirty healthy cooperative children of both sexes who were between 7-9 years and referred to Pediatric Dentistry Department. Two sound teeth without pulpotomy procedure were extracted and subjected to histological procedures to examine the normal pulp tissue and tissue organization (Negative control). The pulpotomy procedure was performed in sixty primary teeth (by split mouth design).
  group I treated with castor oil
  Arms: Castor oil
Drug: Formocresol — Group II treated with formocresol
  Arms: Formocresol

SUMMARY:
The present study was conducted to evaluate and compare pulp response to Castor oil versus Formocresol as Pulpotomy Medicaments in Primary Teeth

ELIGIBILITY:
Inclusion Criteria:

* healthy cooperative children with sound primary canines indicated for extraction for orthodontic reasons

Exclusion Criteria:

* caries primary canines Presence of systemic pathology

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
The degree of pulp inflammation using score. | 2 weeks to 3 months
  The degree of pulp inflammation using scores from 0 to 5 , 0 mean no inflammation ,5 mean abscess formation .
  Measurement the effect of the castor oil as pulp medicament in treated teeth which subjected to decalcification procedure for histological evaluation under light microscope
The presence or absence of dentin chips formation by using scores 0 or 1. | 2 weeks to 3 months
  The presence or absence of dentin chips formation by using scores 0 or 1.
  Measurement the effect of the castor oil as pulp medicament in treated teeth which subjected to decalcification procedure for histological evaluation under light microscope

CONTACTS AND LOCATIONS:
Overall Officials: shomaa Mostafa Hadwa, PHD, Principal Investigator — Tanta University
Locations (1):
- Faculty of dentistry, Tanta, Egypt